CLINICAL TRIAL: NCT02538172
Title: Monitoring of Specific Cytomegalovirus Cell-mediated Immunity (CMV-CMI) for Optimization of Preventive Strategies Against CMV Infection in High-risk Solid-organ Transplant Recipients
Brief Title: Cell-mediated Immunity for Prevention of CMV Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Oriol Manuel, Privat-Docent (PD), University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STCS FUP # 052
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cytomegalovirus Infections
Keywords: Cell-mediated immunity; Antiviral prophylaxis; Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): T-Track® CMV assay Quantiferon-CMV® assays Valganciclovir
  Interventions: Other: T-Track® CMV assay
- Control (Other): T-Track® CMV assay Quantiferon-CMV® assays Valganciclovir
  Interventions: Other: T-Track® CMV assay

INTERVENTIONS:
Other: T-Track® CMV assay
  Other Names: Quantiferon-CMV® assays; Valganciclovir

SUMMARY:
An open-label randomized controlled trial to adapt the duration of antiviral prophylaxis in D+/R- patients and in R+ patients receiving ATG according to the result of the T-Track® CMV assay. Investigators will include kidney and liver transplant recipients. Patients will be randomized during the first month post transplant.

In the interventional arm, while the patient is on antiviral prophylaxis, CMI will be monitored every 4 weeks from the 2nd month after transplant. Measurement of CMV CMI will be done in real time by using the T-Track® CMV assay. The continuation of antiviral prophylaxis will depend on the result of the assay:

* T-Track positive (patient at lower risk): discontinuation of the antiviral drug
* T-Track negative (patient at higher risk): continuation of the antiviral drug until the maximal duration of prophylaxis (3 to 6 months) The standard arm will receive a standard fixed duration of antiviral prophylaxis (3 months for R+ thymoglobulin treated-patients and 6 months for D+/R- patients). Measurement of CMV CMI by both T-Track® CMV and the Quantiferon-CMV® assays will be done at the same time points of the interventional arm, but the result will not be known by the investigators.

After discontinuation of prophylaxis, patients in both arms will be followed for the development of CMV replication at each visit using the local PCR assay and antiviral therapy will be administered in case of CMV infection according to local guidelines.

The co-primary endpoints will be the incidence of CMV disease or antiviral-treated CMV replication during the first 12 months post transplant AND the duration of antiviral prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* Kidney or liver transplantation
* Scheduled to receive CMV antiviral prophylaxis:
* CMV D+/R- patients
* Patients receiving lymphocyte-depleting antibodies (thymoglobulin® or ATG®)

Exclusion Criteria:

* Unable to provide informed consent
* Unable or unwilling to comply with study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2015-10; Primary Completion 2019-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Incidence of CMV infection | one year
Duration of antiviral prophylaxis | one year

SECONDARY OUTCOMES:
Graft survival | one year
Incidence of CMV viremia using standardized measure | one year

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Manuel, MD, Principal Investigator — University of Lausanne Hospitals
Locations (5):
- Switzerland (5):
  - Universität Basel, Basel
  - Universitätsspital Bern, Bern
  - Hopitaux Universitaires de Genève, Geneva
  - Kantonsspital St.Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

REFERENCES:
- [Result] Manuel O, Husain S, Kumar D, Zayas C, Mawhorter S, Levi ME, Kalpoe J, Lisboa L, Ely L, Kaul DR, Schwartz BS, Morris MI, Ison MG, Yen-Lieberman B, Sebastian A, Assi M, Humar A. Assessment of cytomegalovirus-specific cell-mediated immunity for the prediction of cytomegalovirus disease in high-risk solid-organ transplant recipients: a multicenter cohort study. Clin Infect Dis. 2013 Mar;56(6):817-24. doi: 10.1093/cid/cis993. Epub 2012 Nov 29. PMID 23196955
- [Result] Manuel O. Clinical Experience with Immune Monitoring for Cytomegalovirus in Solid-Organ Transplant Recipients. Curr Infect Dis Rep. 2013 Sep 29. doi: 10.1007/s11908-013-0369-6. Online ahead of print. PMID 24078428
- [Result] Humar A, Lebranchu Y, Vincenti F, Blumberg EA, Punch JD, Limaye AP, Abramowicz D, Jardine AG, Voulgari AT, Ives J, Hauser IA, Peeters P. The efficacy and safety of 200 days valganciclovir cytomegalovirus prophylaxis in high-risk kidney transplant recipients. Am J Transplant. 2010 May;10(5):1228-37. doi: 10.1111/j.1600-6143.2010.03074.x. Epub 2010 Mar 26. PMID 20353469
- [Derived] Manuel O, Laager M, Hirzel C, Neofytos D, Walti LN, Hoenger G, Binet I, Schnyder A, Stampf S, Koller M, Mombelli M, Kim MJ, Hoffmann M, Koenig K, Hess C, Burgener AV, Cippa PE, Hubel K, Mueller TF, Sidler D, Dahdal S, Suter-Riniker F, Villard J, Zbinden A, Pantaleo G, Semmo N, Hadaya K, Enriquez N, Meylan PR, Froissart M, Golshayan D, Fehr T, Huynh-Do U, Pascual M, van Delden C, Hirsch HH, Juni P, Mueller NJ; Swiss Transplant Cohort Study (STCS). Immune Monitoring-Guided Versus Fixed Duration of Antiviral Prophylaxis Against Cytomegalovirus in Solid-Organ Transplant Recipients: A Multicenter, Randomized Clinical Trial. Clin Infect Dis. 2024 Feb 17;78(2):312-323. doi: 10.1093/cid/ciad575. PMID 37738676